CLINICAL TRIAL: NCT07352215
Title: Evaluating the Effectiveness of Platelet-Rich Plasma as an Adjunct to Fractional Carbon Dioxide Laser Therapy in Improving Facial Acne Scar Appearance: A Randomized Controlled Trial
Brief Title: PRP Plus Fractional CO₂ Laser for Acne Scars
Acronym: PRPLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gujranwala medical college District Headquarters Hospital, Gujranwala (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Yasaan Saaqib, Principal investigator, Gujranwala medical college District Headquarters Hospital, Gujranwala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: No. IRB.22/ GMC; CPSP/REU/DER-2023-093-19340 (Other: CPSP, Pakistan)
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Post-Acne Atrophic Scars; Carbon Dioxide Lasers; Platelet-Rich Plasma
Keywords: Post-acne Scarring; Fractional CO₂ Laser; PRP Therapy; Skin Resurfacing

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups. One group will receive fractional CO₂ laser combined with platelet-rich plasma (PRP), while the second group will receive fractional CO₂ laser alone. Each participant remains in the same assigned group for the entire study duration, and the interventions are delivered independently and simultaneously across both groups without crossover.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study uses single masking. Participants are blinded to their group assignment by placebo-filled syringes covered with opaque tape applied to the skin without injection to mimic the appearance and procedure of PRP application in control group.
  The treating physician and study staff are aware of the allocation, while the patients and the outcome statistician remain blinded to group identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser + PRP arm (Experimental): Participants receive fractional CO₂ laser treatment followed by the application of autologous platelet-rich plasma (PRP). Three sessions are administered at four-week intervals. PRP is prepared using a double-spin centrifugation method and applied topically immediately after laser treatment.
  Interventions: Procedure: Fractional CO₂ Laser + Platelet-Rich Plasma (PRP)
- Laser only arm (Experimental): Participants receive fractional CO₂ laser treatment alone, without PRP. Three sessions are administered at four-week intervals using the same laser parameters as the intervention group. To maintain masking, a placebo-filled syringe covered with opaque tape is touched to the skin without delivering PRP.
  Interventions: Procedure: Fractional CO₂ Laser Only

INTERVENTIONS:
Procedure: Fractional CO₂ Laser + Platelet-Rich Plasma (PRP) — Fractional CO₂ Laser + Platelet-Rich Plasma (PRP)
  Participants receive fractional CO₂ laser treatment followed by topical application of autologous platelet-rich plasma. Three treatment sessions are performed at four-week intervals. PRP is prepared using a standardized double-spin centrifugation method from 10 mL of the participant's blood. After laser resurfacing, the PRP is applied immediately to the treated area to enhance healing and collagen remodeling.
  Arms: Laser + PRP arm
Procedure: Fractional CO₂ Laser Only — Fractional CO₂ Laser Only
  Participants receive fractional CO₂ laser treatment alone, with the same laser settings and treatment schedule as the intervention group. Three sessions are performed at four-week intervals. To maintain participant blinding, a placebo-filled syringe covered with opaque tape is applied to the skin without delivering PRP.
  Arms: Laser only arm

SUMMARY:
This randomized controlled trial aims to evaluate whether adding platelet-rich plasma (PRP) to fractional CO₂ laser resurfacing improves the treatment of moderate-to-severe acne scars compared with laser alone. Seventy adults aged 18-40 years will be recruited from the Dermatology Department of Gujranwala Medical College Teaching Hospital. Participants will be randomly assigned to receive either fractional CO₂ laser combined with topical PRP or fractional CO₂ laser alone, with three treatment sessions delivered four weeks apart.

The primary outcome is the change in acne scar severity measured using the Goodman and Baron Quantitative Acne Scar Scale. Secondary outcomes include redness, edema, pain scores, and patient satisfaction assessed using Likert and numeric rating scales. The study is single-blinded, with patients unaware of treatment allocation. PRP will be prepared using a standardized double-spin centrifugation process. Data will be analyzed using appropriate statistical tests with a significance level of p < 0.05. The study aims to determine whether PRP enhances laser efficacy, reduces side effects, and improves patient-reported outcomes.

DETAILED DESCRIPTION:
Acne scarring is a frequent and distressing outcome of acne vulgaris. Fractional carbon dioxide (CO₂) laser therapy is widely used for acne scar management because it creates controlled microthermal zones that stimulate collagen remodeling and improve skin texture. However, laser treatment alone may lead to side effects such as erythema, edema, discomfort, and variable degrees of clinical improvement.

Platelet-rich plasma (PRP) is an autologous biological product containing high concentrations of platelets, growth factors, and cytokines known to promote wound healing, enhance collagen production, and modulate inflammation. The combination of PRP with fractional CO₂ laser treatment is believed to enhance clinical results, improve healing time, and reduce post-procedural complications. This study is designed to evaluate whether adding PRP to fractional CO₂ laser improves outcomes for patients with moderate-to-severe acne scars.

This randomized controlled trial will recruit 70 patients aged 18-40 years with moderate-to-severe facial acne scars. Participants will be randomly allocated into two groups. Group A will receive fractional CO₂ laser therapy combined with PRP, and Group B will receive fractional CO₂ laser therapy alone. Both groups will undergo three treatment sessions spaced four weeks apart. The study uses single blinding, where patients are unaware of their treatment assignment. To maintain blinding, a placebo-filled syringe will be used in the control group and gently applied without injecting any substance.

PRP will be prepared using a standardized double-spin method. Ten milliliters of venous blood will be collected in anticoagulant tubes, centrifuged at low speed to separate plasma and buffy coat, followed by a second high-speed centrifugation to isolate platelet-rich plasma. Topical anesthesia with lignocaine-prilocaine cream will be applied before each laser session. Treatment areas will be prepared using antiseptic measures, and eye protection will be provided.

Outcome assessment will be performed at baseline and at each visit. The primary outcome is the change in acne scar severity measured using the Goodman and Baron Quantitative Acne Scar Scale. Secondary outcomes include assessments of erythema and edema by the evaluator, as well as patient-reported pain scores and satisfaction ratings. Standardized clinical photographs will support patient self-assessment under consistent lighting and camera settings.

Data will be analyzed using appropriate statistical methods. Continuous variables will be assessed for normality and compared using t-tests or nonparametric equivalents. Categorical and ordinal data will be analyzed using Chi-square or related tests. A significance level of p < 0.05 will be applied. Data will be coded, and the statistician will remain blinded to group allocation.

The purpose of this trial is to determine whether PRP enhances the efficacy, safety profile, and patient satisfaction of fractional CO₂ laser treatments. If successful, this combination approach may offer a more effective therapeutic option for managing moderate-to-severe acne scarring.

ELIGIBILITY:
Inclusion Criteria:Adults aged 18 to 40 years

Male and female participants

Fitzpatrick skin types I to V

Presence of moderate-to-severe acne scars

Willing to undergo 3 treatment sessions and follow-up visits

Able to provide informed consent -

Exclusion Criteria:Use of topical anti-acne medications in the past 1 month

History of keloid formation or hypertrophic scarring

Active acne or active skin inflammation at treatment area

Diabetes mellitus

Photosensitive disorders (e.g., lupus, dermatomyositis)

Melasma

Active infections (e.g., Herpes simplex)

Recent laser resurfacing or similar procedures

Outdoor workers with high sun exposure

Vitiligo

Pregnancy or breastfeeding

Bleeding disorders or anticoagulant therapy

Unrealistic expectations or inability to comply with follow-up

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Acne Scar Severity (Goodman and Baron Quantitative Acne Scar Scale) | 12weeks
  Acne scar severity will be assessed using the Goodman and Baron Quantitative Acne Scar Scale, which grades scars based on type, number of lesions, and affected surface area. Scores will be recorded at baseline and at each follow-up visit to measure improvement over the course of treatment.

SECONDARY OUTCOMES:
Redness (Erythema) Score | 12weeks
  Redness will be evaluated by the assessor using a 4-point Likert scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) at each visit to assess post-laser inflammatory response.
Edema (Swelling) Score | 12 weeks
  Edema will be assessed by the evaluator using a 4-point Likert scale ranging from 0 (none) to 3 (severe) to evaluate treatment-related swelling.
Pain Score (11-Point Numeric Rating Scale) | 12 weeks
  Participants will report pain intensity using an 11-point numeric scale (0 = no pain; 10 = worst possible pain) during and after each treatment session.
Patient Satisfaction Rating | 12 weeks
  Patient satisfaction with treatment outcome will be measured using a 4-point Likert scale (0 = not satisfied; 1 = neutral; 2 = satisfied; 3 = very satisfied). Standardized digital photographs will be used to assist patient self-evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: YASAAN SAAQIB, Principal Investigator — Gujranwala Medial College Gujranwala
Locations (1):
- Destrict Head Quarter Hospital, Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
I sill do it after publication of my study

REFERENCES:
- [Background] Rullan PP, Olson R, Lee KC. A Combination Approach to Treating Acne Scars in All Skin Types: Carbolic Chemical Reconstruction of Skin Scars, Blunt Bi-level Cannula Subcision, and Microneedling-A Case Series. J Clin Aesthet Dermatol. 2020 May;13(5):19-23. Epub 2020 May 1. PMID 32802250
- [Result] Connolly D, Vu HL, Mariwalla K, Saedi N. Acne Scarring-Pathogenesis, Evaluation, and Treatment Options. J Clin Aesthet Dermatol. 2017 Sep;10(9):12-23. Epub 2017 Sep 1. PMID 29344322